CLINICAL TRIAL: NCT02774044
Title: Evaluating the Efficacy and Safety of an Innovative and Affordable Goat Lung Surfactant for the Treatment of Respiratory Distress Syndrome in Preterm Neonates: a Multi-site Randomized Clinical Trial
Brief Title: Efficacy and Safety of Goat Lung Surfactant for the Treatment of Respiratory Distress Syndrome in Preterm Neonates
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ramesh K Agarwal (Other)
Collaborators: Maulana Azad Medical College, New Delhi (Unknown); Lady Hardinge Medical College (Other Government); Chacha Nehru Bal Chikitsalya, Delhi (Unknown); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); King Edward Memorial Hospital, Mumbai (Other Government); Lokmanya Tilak Municipal General Hospital, Mumbai (Unknown); Institute of Child health and Hospital for Children, Chennai (Unknown); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); All India Institute of Medical Sciences (Other); St Johns Medical College Hospital, Bangalore, India (Other); King Edward Memorial Hospital, Pune (Unknown); Government Medical College, Chandigarh (Other); Wellcome Trust (Other)
Responsible Party: Sponsor-Investigator, Ramesh K Agarwal, Additional Professor, All India Institute of Medical Sciences
Organization: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N1617
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: preterm neonates, surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — goat lung surfactant extract; beractant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cadisurf (goat lung surfactant extract) (Experimental): Neonates in the intervention group will be intratracheally administered 100 mg/kg of GLSE (CADISURF®).
  Interventions: Drug: Cadisurf
- Survanta (Beractant) (Active Comparator)
  Interventions: Drug: Survanta

INTERVENTIONS:
Drug: Cadisurf — Cadisurf Intratracheal suspension is a sterile, non-pyrogenic pulmonary surfactant intended for intratracheal use only. It is a natural lung extract containing phospholipids and surfactant-associated proteins. The resulting composition provides 25 mg/mL phospholipids and less than 1.0 mg/ml protein. It is suspended in 0.9% sodium chloride solution. Cadisurf contains no preservatives. Each ml of Cadisurf contains 25 mg of phospholipids. It is a creamy white suspension supplied in single-use glass vials containing 8 mL (200 mg phospholipids).
  Other Names: Goat lung surfactant extract
  Arms: Cadisurf (goat lung surfactant extract)
Drug: Survanta
  Other Names: Beractant
  Arms: Survanta (Beractant)

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Cadisurf (goat lung surfactant extract) as compared to Survanta (beractant) in the treatment of respiratory distress syndrome in preterm neonates (with gestation of 26 to 32 weeks).

DETAILED DESCRIPTION:
Title: Evaluating the Efficacy and Safety of an Innovative and Affordable Lung Surfactant for the treatment of Respiratory Distress Syndrome (RDS) in preterm neonates: a multi-site randomized clinical trial

Phase of Development: Phase II/ III

Indication: Respiratory Distress Syndrome

Primary Objective: To compare the incidence of survival without bronchopulmonary dysplasia (BPD) at 36 weeks postmenstrual age in preterm neonates (≤32 wk) with RDS randomized to receive intratracheal administration (100 mg/kg) of either goat lung surfactant extract (GLSE) or the standard preparation (Beractant; Survanta; Abbott, USA)

Secondary Objective: 1 To compare area under curve (AUC) for oxygen requirement (FiO2) requirement in first 48 h of surfactant administration

2 To compare incidence of safety outcomes namely air leaks, pulmonary hemorrhage, intraventricular hemorrhage, neonatal mortality, sepsis and retinopathy of prematurity

Study Design: A multicentric, non-inferiority randomized controlled trial (RCT) in preterm infants with RDS.

Study Centers: The study would be conducted at 12-14 academic centers of India.

Study population: A total of approximately 900 eligible preterm neonates will be enrolled in the study.

Planned No. of subjects: N~900 to be enrolled by 12-14 centers

Investigational Product : GLSE (Lung Surfactant Extract) Cadisurf 25

Dosage and site of administration: Dosage: Neonates in the intervention group will be administered 100 mg/kg of GLSE. Those in the control group will be administered 100 mg/kg of Beractant (Survanta®, Abbott, USA).

Site of Administration: Intratracheal

Expected Duration of Participation of each Subject: 4-10 Weeks

Expected duration of study 3 years

Methodology The study would be conducted at 12-14 study sites. The dedicated study teams under the leadership of site Principal Investigator (PI) at each site would implement the study protocol as per uniform standard operating procedures (SOPs). Written informed consent will be taken from the legally authorized representative (LAR) of the subject. Subjects will be enrolled based on the inclusion/exclusion criteria depicted in the institute ethics committee (IEC) & Central drugs standard control organization (CDSCO) approved protocol. After satisfying inclusion/exclusion criteria subjects will be randomized either GLSE arm or Beractant (Survanta®, Abbott, USA) arm. The duration of the hospitalization would be 4-10 weeks. Enrolled infants would be monitored by the study team round the clock as per standard procedures. The study infants would be followed up until death or 36 weeks of postmenstrual age (PMA). Adverse events & serious adverse events will be recorded & reported as per the regulatory guidelines of India.

The study infants would be followed up until 36 weeks of PMA. The study would be conducted at 12-14 study sites. The study will be conducted in a highly supervised clinical setting with immediate availability of clinicians experienced with intubation, ventilator management and general care of premature infants. Infants receiving surfactant will be frequently monitored with arterial or transcutaneous measurement of systemic O2 and CO2. The dedicated study teams at each site would implement the study protocol as per uniform standard operating procedures (SOPs).

Primary Study Endpoint • BPD free survival

Blinding Procedures

1. Random sequence The random sequence will be generated using web based algorithm for 1:1 allocation and stratification by site and gestation (<28 and 28-32 weeks) in permuted blocks of random sizes. The block sizes will be blinded to the investigators.
2. Allocation concealment The vials of two surfactant products would be packaged in identical cardboard boxes (by CDSA) and sequentially numbered as per the allocation sequence for two gestation strata (8 mL vials for strata 26-27 weeks and 28-32 weeks, respectively) for each site.
3. Implementation The randomization sequence would be generated by an independent statistician and will be kept in safe custody and undisclosed to investigators.

   Dedicated research teams would track, ascertain the eligibility and randomize the infants and measure the outcomes. The clinical team would administer surfactant blinded to research team.
4. Blinding Clinicians would be aware of the type of surfactant product received by the neonate given the different physical appearance of the product and the vial of Cadisurf® and Survanta®. Clinicians would administer the surfactant to the baby while the baby's bed is cordoned off from rest of NICU by cloth screen. The parents and the research staff responsible for outcome assessment would be kept blinded to the interventions. The allocation would be concealed in the dataset so that the researchers can analyse data without information of the allocation.

Interim analysis Interim analyses, if desired by the Data Safety Monitoring Board (DSMB), are proposed at enrolment of 5%, 33% and 66% of the target sample size. The DSMB would only have access to the results of such analyses. Interim analysis will be conducted using O'Brien-Fleming spending function and a type I error rate of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at the study sites and fulfilling all of the following criteria will be eligible for enrolment in the study

  1. Gestational age ≤32 completed weeks
  2. Onset of respiratory distress within six hours of age
  3. If baby meets criteria for surfactant replacement therapy:

     1. FiO2 needed is 40% or higher while the baby is on CPAP to maintain pre-ductal oxygen saturation between 90% to 95% or
     2. Baby needs intubation because of CPAP failure or severe respiratory distress (Chest X-ray is not mandatory for deciding the need for SRT). Detailed SOPs will be developed with respect to assessing the eligibility for SRT

        Exclusion Criteria:

        Neonates with any of the following criteria will be excluded:

  <!-- -->

  1. Gestation below 26 wk
  2. Babies with severe birth asphyxia as defined by the need for chest compressions and/or initial (umbilical arterial/or within 1 hour of birth) pH <7.0
  3. Major congenital malformations
  4. Prophylactic surfactant administration, i.e. administration of surfactant before the infant develops respiratory distress
  5. Air leak or pulmonary hemorrhage prior to enrollment
  6. Shock requiring vasopressor support prior to enrollment

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
BPD free survival | 36 weeks post menstrual age
  Survival free from BPD defined as per the definition provided by NIH

SECONDARY OUTCOMES:
Area under the curve for (AUC) for oxygen requirement (FiO2) requirement in first 48 h | 48 hours after surfactant replacement therapy
  The oxygen requirement will be recorded every hour using a standardized protocol and AUC for first 48 hrs will be calculated. The outcome would be recorded by the study staff and AUC calculated in a subset of 250 infants.
Pulmonary haemorrhage | 48 hours after surfactant replacement therapy
  Occurrence of bleeding/blood stained secretions from the trachea within 48 hr of surfactant administration
Any air leak within 72 hours of administration of surfactant | 72 hours after surfactant replacement therapy
  Occurrence of any airleak -pneumothorax, PIE or pneumomediastinum in chest X-ray (done when clinically suspected)
IVH grade 3 or 4 | 72±24 hrs
  Grade 3 or 4 IVH as per Papille/Volpe classification
Periventricular Leukomalacia (PVL)-cystic and non-cystic | 72±24 hrs
  PVL as per deVries classification
PVL-cystic and non-cystic | 28±7days
  PVL as per deVries classification
Sepsis | 7 days of age
  Occurrence of any episode of sepsis (culture positive or culture negative) from the time of enrolment until 7 days of age
Respiratory support at 72 h | 72 hours of age
  Mechanical ventilation/CPAP/HFNC/free flow oxygen/none at the two time points (point assessments)
Respiratory support at 7 days of age | 7 days of age
  Mechanical ventilation/CPAP/HFNC/free flow oxygen/none at the two time points (point assessments)
Retinopathy of prematurity (ROP) | Eyes of the babies would be examined by the ophthalmologists starting from 4 wk of life
  ROP requiring laser as per ICROP classification
Neonatal Mortality | first 28 days of life
  Death of a neonate in first 28 days of life
Duration of mechanical ventilation and CPAP | 36 weeks postmenstrual age
  Cumulative duration of mechanical ventilation and CPAP until discharge/death
Duration of hospital stay | 36 weeks postmenstrual age
  Duration of hospital stay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jain K, Nangia S, Ballambattu VB, Sundaram V, Sankar MJ, Ramji S, Vishnubhatla S, Thukral A, Gupta YK, Plakkal N, Sundaram M, Jajoo M, Kumar P, Jayaraman K, Jain A, Saili A, Murugesan A, Chawla D, Murki S, Nanavati R, Rao S, Vaidya U, Mehta A, Arora K, Mondkar J, Arya S, Bahl M, Utture A, Manerkar S, Bhat SR, Parikh T, Kumar M, Bajpai A, Sivanandan S, Dhawan PK, Vishwakarma G, Bangera S, Kumar S, Gopalakrishnan S, Jindal A, Natarajan CK, Saini A, Karunanidhi S, Malik M, Narang P, Kaur G, Yadav CP, Deorari A, Paul VK, Agarwal R. Goat lung surfactant for treatment of respiratory distress syndrome among preterm neonates: a multi-site randomized non-inferiority trial. J Perinatol. 2019 Sep;39(Suppl 1):3-12. doi: 10.1038/s41372-019-0472-0. PMID 31485014